CLINICAL TRIAL: NCT05795933
Title: Efficacy of Vitamin D Supplementation for Children With Bronchiolitis at Sohag University Hospital
Brief Title: Efficacy of Vitamin D Supplementation for Children With Bronchiolitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Youstina Safwat Labib, Pediatric Resident, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-03-11MS
Record Dates: First submitted 2023-03-08; First posted 2023-04-03 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; Vitamin D; Children
MeSH Terms: conditions — Bronchiolitis | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Two groups of children with bronchiolitis:
  Study group: will receive a single dose of intramuscular 200,000 IU vitamin D3 within 24 hours of admission.
  Control group: will receive the standard recommended dose of vitamin D3 as 400 IU/day orally
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Children receive a single dose of intramuscular 200,000 IU vitamin D3
  Interventions: Drug: Vitamin D3
- Control group (No Intervention): Children receiving only the standard recommended dose of vitamin D3 as 400 IU/day orally

INTERVENTIONS:
Drug: Vitamin D3 — A single dose of intramuscular 200,000 IU vitamin D3 within 24 hours of admission
  Other Names: Cholecalciferol; Devarol
  Arms: Study group

SUMMARY:
Vitamin D plays an important role in enhancing mucosal immune defense, decreasing excessive inflammation, and increasing mucociliary clearance. Experimental studies have shown that vitamin D reduces inflammation of epithelial cells in airways infected with Respiratory Syncytial Virus and confers antiviral effects. Furthermore, several studies have shown lower serum vitamin D levels in hospitalized children with bronchiolitis. However, studies on the efficacy of Vitamin D supplementation for children with bronchiolitis are scarce with inconsistent findings. In this study, we aim to evaluate the efficacy of vitamin D supplementation in children with bronchiolitis.

DETAILED DESCRIPTION:
Bronchiolitis is the most frequent lower respiratory tract infection in children under two years of age, which represents a major cause of medical visits, hospital admissions, and death. This disease predominantly affects small airways with acute inflammatory edema epithelial cells, excess mucus production, and bronchospasm. The most commonly involved organisms are Respiratory Syncytial Virus (accounting for 60% of cases), followed by Rhinovirus, Parainfluenza, Metapneumovirus, Influenza, and Adenovirus. Certain factors are associated with a higher risk of severe bronchiolitis, such as prematurity, chronic lung disease, cardiac disease, immunodeficiency, neuromuscular disease, and Down syndrome.

Diagnosis of bronchiolitis relies on a constellation of clinical manifestations, including respiratory distress and wheezing preceded by viral upper respiratory tract prodrome in children under two years of age. Common manifestations of bronchiolitis are rhinorrhea, cough, wheezing, tachypnea, and increased work of breathing, including nasal flaring, retractions, and grunting. Management of bronchiolitis is mainly supportive, aiming at maintaining adequate oxygenation and hydration.

Given the high burden of bronchiolitis and the lack of specific treatment, studies have investigated several therapeutic options. One of these potential therapies is vitamin D. Vitamin D is a fat-soluble vitamin that is mainly formed in the skin after exposure to ultraviolet rays, while less than 10% is obtained from dietary sources. Besides regulation of calcium and phosphorus homeostasis, vitamin D plays an important role in enhancing mucosal immune defense, decreasing excessive inflammation, and increasing mucociliary clearance. Vitamin D deficiency is common among children, particularly in developing countries, and has been linked to an increased risk of several diseases, including bronchiolitis, pneumonia, and otitis media.

Experimental studies have shown that vitamin D reduces inflammation of epithelial cells in airways infected with Respiratory Syncytial Virus and confers antiviral effects. Furthermore, several studies have shown lower serum vitamin D levels in hospitalized children with bronchiolitis. However, studies on the efficacy of Vitamin D supplementation for children with bronchiolitis are scarce with inconsistent findings.

In this study, we aim to evaluate the efficacy of vitamin D supplementation in children with bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 to 24 months.
* Clinical diagnosis of first episode of bronchiolitis
* First 24 hours of admission.
* Stable or decreasing requirement for oxygen on 2 measurements 2 hours apart.
* Pulse rate less than 180 beat/minute.
* Respiratory rate less than 80 breath/min.
* Oxygen supplementation < 40% Fraction of inspired oxygen or < 2 L/min by nasal prong
* Not on high flow nasal cannula, continuous positive airway pressure, or mechanical ventilation at the time of enrollment.

Exclusion Criteria:

.• History of previous episodes of wheezing.

* History of apnea
* Need for positive pressure support or high flow nasal cannula at the time of enrollment.
* Chronic lung disease (requiring home oxygen, or pulmonary hypertension)
* Cardiac disease (cyanotic, hemodynamically significant [requiring diuretics], or pulmonary hypertension).
* Neuromuscular disease.
* Metabolic disease.
* Immunodeficiency.
* Chromosomal abnormalities.
* Craniofacial malformation
* Hemoglobinopathy.
* Hypercalcemia
* Chromosomal abnormalities
* Use of large doses of vitamin D (> 400 IU/day) in the last month.

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
Time from randomization to discharge | 4 weeks
  Time from randomization to hospital discharge (in hours)

SECONDARY OUTCOMES:
Time from randomization to discontinuation of oxygen therapy | 4 weeks
  Time from randomization to discontinuation of oxygen therapy (in hours)
Time from randomization to discontinuation of intravenous fluids | 4 weeks
  Time from randomization to discontinuation of intravenous fluids (in hours)
Time from randomization to meeting discharge criteria | 4 weeks
  Time from randomization to meeting hospital discharge criteria (in hours)
Time from hospital admission to discharge | 4 weeks
  Time from hospital admission to discharge (in hours)
Blood level of 25-hydroxycholecalciferol | On day 3 after randomization
  Blood level of 25-hydroxycholecalciferol
Serum level of ionized calcium | On day 3 after randomization
  Serum level of ionized calcium
Admission to pediatric intensive care unit | 4 weeks
  Proportion of patients admitted to pediatric intensive care unit
Intubation | 4 weeks
  Proportion of patients who underwent endotracheal intubation
Mortality | 4 weeks
  Proportion of patients who died during hospital admission
Bronchodilator therapy | 4 weeks
  Proportion of patients who received bronchodilator therapy
Systemic steroids | 4 weeks
  Proportion of patients who received systemic steroids

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa A Mohammed, MD, PhD, Study Chair — Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Unidentified patients' data will be available upon reasonable request after publication
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the study
Access Criteria: Unidentified patients' data will be available upon reasonable request after publication

REFERENCES:
- [Background] Manti S, Staiano A, Orfeo L, Midulla F, Marseglia GL, Ghizzi C, Zampogna S, Carnielli VP, Favilli S, Ruggieri M, Perri D, Di Mauro G, Gattinara GC, D'Avino A, Becherucci P, Prete A, Zampino G, Lanari M, Biban P, Manzoni P, Esposito S, Corsello G, Baraldi E. UPDATE - 2022 Italian guidelines on the management of bronchiolitis in infants. Ital J Pediatr. 2023 Feb 10;49(1):19. doi: 10.1186/s13052-022-01392-6. PMID 36765418
- [Background] Ralston SL, Lieberthal AS, Meissner HC, Alverson BK, Baley JE, Gadomski AM, Johnson DW, Light MJ, Maraqa NF, Mendonca EA, Phelan KJ, Zorc JJ, Stanko-Lopp D, Brown MA, Nathanson I, Rosenblum E, Sayles S 3rd, Hernandez-Cancio S; American Academy of Pediatrics. Clinical practice guideline: the diagnosis, management, and prevention of bronchiolitis. Pediatrics. 2014 Nov;134(5):e1474-502. doi: 10.1542/peds.2014-2742. PMID 25349312
- [Background] Munns CF, Shaw N, Kiely M, Specker BL, Thacher TD, Ozono K, Michigami T, Tiosano D, Mughal MZ, Makitie O, Ramos-Abad L, Ward L, DiMeglio LA, Atapattu N, Cassinelli H, Braegger C, Pettifor JM, Seth A, Idris HW, Bhatia V, Fu J, Goldberg G, Savendahl L, Khadgawat R, Pludowski P, Maddock J, Hypponen E, Oduwole A, Frew E, Aguiar M, Tulchinsky T, Butler G, Hogler W. Global Consensus Recommendations on Prevention and Management of Nutritional Rickets. J Clin Endocrinol Metab. 2016 Feb;101(2):394-415. doi: 10.1210/jc.2015-2175. Epub 2016 Jan 8. PMID 26745253
- [Background] Esposito S, Lelii M. Vitamin D and respiratory tract infections in childhood. BMC Infect Dis. 2015 Oct 28;15:487. doi: 10.1186/s12879-015-1196-1. PMID 26521023
- [Background] Golan-Tripto I, Loewenthal N, Tal A, Dizitzer Y, Baumfeld Y, Goldbart A. Vitamin D deficiency in children with acute bronchiolitis: a prospective cross-sectional case- control study. BMC Pediatr. 2021 Apr 30;21(1):211. doi: 10.1186/s12887-021-02666-4. PMID 33931018
- [Background] Khoshnevisasl P, Sadeghzadeh M, Kamali K, Ardalani A. A randomized clinical trial to assess the effect of zinc and vitamin D supplementation in addition to hypertonic saline on treatment of acute bronchiolitis. BMC Infect Dis. 2022 Jun 13;22(1):538. doi: 10.1186/s12879-022-07492-2. PMID 35692038
- [Background] Wang EE, Milner RA, Navas L, Maj H. Observer agreement for respiratory signs and oximetry in infants hospitalized with lower respiratory infections. Am Rev Respir Dis. 1992 Jan;145(1):106-9. doi: 10.1164/ajrccm/145.1.106. PMID 1731571
- [Background] Brustad N, Yousef S, Stokholm J, Bonnelykke K, Bisgaard H, Chawes BL. Safety of High-Dose Vitamin D Supplementation Among Children Aged 0 to 6 Years: A Systematic Review and Meta-analysis. JAMA Netw Open. 2022 Apr 1;5(4):e227410. doi: 10.1001/jamanetworkopen.2022.7410. PMID 35420658
- [Background] Sarhan AA, Saeed NM, Mostafa AA, Osman AM. Vitamin D supplementation for acute bronchiolitis: a double-blind randomized controlled trial. Alexandria Journal of Pediatrics. 2019;32(2):61.
- [Background] Saad K, Abd Aziz NH, El-Houfey AA, El-Asheer O, Mohamed SA, Ahmed AE, Abdel Baseer KA, Darwish MM. Trial of vitamin D supplementation in infants with bronchiolitis: a randomized, double-blind, placebo-controlled study. Pediatric Allergy, Immunology, and Pulmonology. 2015;28(2):102-6